CLINICAL TRIAL: NCT06644183
Title: A Phase 1/2, Open Label, Study of Roginolisib (IOA-244), an Orally Bioavailable, Selective PI3Kδ Inhibitor in Patients With Refractory/Relapsed Chronic Lymphocytic Leukemia (CLL) in Combination With Venetoclax and Rituximab
Brief Title: Roginolisib (IOA-244) With Venetoclax and Rituximab for Refractory/Relapsed Chronic Lymphocytic Leukemia (CLL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jennifer R. Brown, MD, PhD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jennifer R. Brown, MD, PhD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-449
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Leukemia; Relapsed Leukemia; Chronic Lymphocytic Leukemia; Relapsed Cancer; Refractory Leukemia
Keywords: Leukemia; Relapsed Leukemia; Chronic Lymphocytic Leukemia; Relapsed Cancer; Refractory Leukemia; CLL; Relapsed Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — venetoclax; Rituximab

STUDY DESIGN:
Intervention Model Description: Phase 1: single arm, Phase 2: two arm, randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b Arm A: Venetoclax + Roginolisib + Rituximab Dose Level -1 (Experimental): 3+3 design to establish a Recommended Phase 2 Dose (RP2D) for Roginolisib, starting at Dose Level -1.
  * Baseline visit, imaging, bone marrow biopsy
  * CT scan every 2 cycles
  * Cycle 1 (5 weeks): Predetermined dose of Venetoclax 1x daily
  * Cycle 2: Days 1 through 28 of 28 day cycle: Predetermined dose of Venetoclax 1x daily and predetermined dose of Roginolisib 1 x daily
    --If 0 of 3 participants do not experience a dose-limiting toxicity (DLT), the study will proceed. If 1 of 3 participants experience a DLT, 3 more participants will be enrolled, and if 1 of those 6 participants experience a DLT, this is the RP2D for phase 2. If a DLT is observed in 2 of 3 or 2 of 6, the study will be stopped.
  * Cycles 3 through Cycle 8: Day 1 of 28 day cycle: Predetermined dose of Rituximab once
  * Cycles 3 through 13: Days 1 through 28 of 28 day cycle: Predetermined dose of Venetoclax 1x daily and predetermined dose of Roginolisib 1 x daily
  * End of treatment visit
  * Follow up visits for up to 5 years
  Interventions: Drug: Roginolisib; Drug: Venetoclax; Drug: Rituximab
- Phase 1b Arm B: Venetoclax + Roginolisib + Rituximab Dose Level 1 (Experimental): * Baseline visit, imaging, bone marrow biopsy
  * CT scan every 2 cycles
  * Cycle 1 (5 weeks): Predetermined dose of Venetoclax 1x daily
  * Cycle 2: Days 1 through 28 of 28 day cycle: Predetermined dose of Venetoclax 1x daily and predetermined dose of Roginolisib 1 x daily
    --If 0 of 3 participants do not experience a DLT, Phase 2 will start at this dose level. If 1 of 3 participants experience a DLT, 3 more participants will be enrolled, and if 1 of those 6 participants experience a DLT, this dose level will be used for Phase 2. If a DLT is observed in 2 of those 6, de-escalate to Dose Level -1.
  * Cycles 3 through Cycle 8: Day 1 of 28 day cycle: Predetermined dose of Rituximab once
  * Cycles 3 through 13: Days 1 through 28 of 28 day cycle: Predetermined dose of Venetoclax 1x daily and predetermined dose of Roginolisib 1 x daily
  * End of treatment visit
  * Follow up visits for up to 5 years
  Interventions: Drug: Roginolisib; Drug: Venetoclax; Drug: Rituximab
- Phase 2 Arm A: Venetoclax + Roginolisib + Rituximab (Experimental): Participants will be randomized 1:1 and stratified by TP53 aberrant disease and by the number of prior therapies.
  * Baseline visit, imaging, bone marrow biopsy.
  * CT scan every 2 cycles.
  * Cycle 1 (5 weeks): Predetermined dose of Venetoclax 1x daily
  * Cycles 2 through 13:
    * Days 1 through 28 of 28 day cycle: Predetermined dose of Venetoclax 1x daily.
    * Days 1 through 28 of 28 day cycle: Predetermined dose of Roginolisib 1 x daily.
  * Cycles 3 through Cycle 8:
    --Day 1 of 28 day cycle: Predetermined dose of Rituximab once.
  * End of treatment visit
  * Follow up visits for up to 5 years
  Interventions: Drug: Roginolisib; Drug: Venetoclax; Drug: Rituximab
- Phase 2 Arm B: Venetoclax + Rituximab (Active Comparator): Participants will be randomized 1:1 and stratified by TP53 aberrant disease and by the number of prior therapies.
  * Baseline visit, imaging, bone marrow biopsy.
  * CT scan every 2 cycles.
  * Cycle 1 (5 weeks): Predetermined dose of Venetoclax 1x daily
  * Cycles 2 through 13:
    --Days 1 through 28 of 28 day cycle: Predetermined dose of Venetoclax 1x daily.
  * Cycle 3 through 8:
    --Day 1 of 28 day cycle: Predetermined dose of Rituximab once.
  * End of treatment visit
  * Follow up visits for up to 5 years
  Interventions: Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Roginolisib — Phosphoinositide 3-kinase delta inhibitor, 40 mg capsule, taken orally per protocol.
  Other Names: MSC2360844A; [6-fluoro-1-(4-morpholin-4-ylmethyl-phenyl)-5,5-dioxo-4,5-dihydro-1H-5λ6-thiochro-meno[4,3-c]pyrazol-3-yl]-morpholin-4-yl-methanone hemi-fumarate, C26 H27 F N4 O5 S. 0.5 C4H4O4
  Arms: Phase 1b Arm A: Venetoclax + Roginolisib + Rituximab Dose Level -1; Phase 1b Arm B: Venetoclax + Roginolisib + Rituximab Dose Level 1; Phase 2 Arm A: Venetoclax + Roginolisib + Rituximab
Drug: Venetoclax — B-cell lymphoma 2 inhibitor, 10, 50, and 100mg tablets, taken orally per standard of care.
  Other Names: ABT-199; GDC-0199
Drug: Rituximab — Chimeric anti-CD 20 monoclonal antibody, single-use 10 and 50mL vials, via intravenous (into the vein) infusion per standard of care.
  Other Names: Riabni; Ruxience; Truxima; Rituxan; ABP 798; IDEC-C2B8, PF-05280586; MabThera

SUMMARY:
This research study will test the safety and anticancer activity of the combination of three drugs (Roginolisib, Venetoclax, and Rituximab) for participants with relapsed or refractory Chronic Lymphocytic Leukemia (CLL).

The names of the study drugs involved in this study are:

* Roginolisib (a novel type of PI3-kinase delta inhibitor)
* Venetoclax (a type of B-cell lymphoma 2 inhibitor)
* Rituximab (a type of monoclonal antibody)

DETAILED DESCRIPTION:
This is a Phase I/II, open-label, randomized, and comparator controlled study to test the safety and anticancer activity of the combination of three drugs (Roginolisib, Venetoclax, and Rituximab) for participants with relapsed or refractory Chronic Lymphocytic Leukemia (CLL). In this study, investigators are assessing whether adding the study drug, Roginolisib, will lead to deeper responses than the standard combination of Venetoclax and Rituximab alone.

A phase Ib safety lead-in portion of the trial will determine the dose and tolerability of Roginolisib with the standard 2-drug combination treatment of Venetoclax + Rituximab.

In the phase 2 portion of the trial, participants will be randomized into one of two treatment arms: Arm A: Roginolisib + Venetoclax and Rituximab vs. Arm B: Venetoclax and Rituximab. Randomization means a participant is placed into a treatment arm by chance.

The U.S. Food and Drug Administration (FDA) has not approved Roginolisib as a treatment for relapsed or refractory CLL.

The U.S. FDA has approved Venetoclax and Rituximab as a standard 2-drug combination treatment for relapsed or refractory CLL.

The research study procedures include screening for eligibility in-clinic visits, blood tests, urine tests, electrocardiograms (ECGs), Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, and bone marrow biopsy and/or aspirations.

Participants will receive study treatment for approximately 12 months and will be followed for up to 5 years.

It is expected about 3-12 people will take part in the Phase 1 portion of the trial, and 52 people will participate in the Phase 2 portion of the research study.

iOnctura SA is supporting this research study by providing the study drug, Roginolisib.

The U.S. Department of Defense (DOD) is supporting this research study by providing funding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory CLL who meet iwCLL criteria for requiring treatment.
* Patients with measurable disease as defined by at least one of: circulating lymphocytosis > 5000 B cells/microliter, bone marrow involvement > 30%, palpable splenomegaly or lymph nodes > 1.5 cm. Computer tomography (CT) at screening must be performed and followed every 2 cycles (1 cycle = 28 days).
* Patients must have received at least two prior therapies for CLL including systemic therapy containing a covalent BTK inhibitor.
* Patients willing to undergo a pre-treatment and on treatment bone marrow biopsy.
* Age ≥18 years, at the time of signing the IRB approved informed consent. Because no dosing or adverse event data are currently available on the use of venetoclax in combination with roginolisib in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Participants must meet the following organ and marrow function as defined below:

  * Platelet count ≥50 x 109/L^^^
  * Total bilirubin ≤ 1.5 ×institutional upper limit of normal (ULN)*
  * AST(SGOT)/ALT(SGPT) ≤3.0 × institutional ULN
  * Creatinine clearance ≥ 60 mL/min**
  * ^^^Thrombocytopenia due to marrow involvement of CLL: > 30 x 109/L for the safety run-in, and 20 x 109/L for the randomized portion of the study
  * *unless increase attributed to leukemic organ involvement, hemolysis or Gilbert's syndrome. Patients who are < 75 years may have bilirubin of ≤ 3.0 × ULN
  * ** calculated by the Cockcroft Gault formula or measured by 24 hours urine collection
* Patients with clinically inactive CNS disease or treated CNS disease that is no longer symptomatic, or who need corticosteroids or anticonvulsants may be enrolled in the study. For patients who have symptoms present, imaging and lumbar puncture must be performed to exclude a CNS condition that may impact the study conduct.
* Willingness to undergo a pre-treatment and on-treatment bone marrow to evaluate MRD.
* Willingness to use adequate contraception prior to study entry and for the duration of study participation.

  * The effects of roginolisib on the developing human fetus are unknown.
  * Venetoclax may cause embryo fetal harm when administered to pregnant women. Anti-CD20 targeting agents are likely to cause fetal B-cell depletion. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women of child-bearing potential will be required to have a negative serum pregnancy test during screening and a negative serum pregnancy test on Cycle 1 Day 1. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of roginolisib or venetoclax administration. Contraception must be conducted up to 12 months after taking the last rituximab dose.
* Ability to understand and the willingness to sign a written informed consent document, which includes compliance with the requirements of this protocol.
* Eligible to receive infection prophylaxis and supportive care as per institutional guidelines.

Exclusion Criteria:

* Patients who have received prior treatment with venetoclax or PI3K inhibitors in the last 6 months. Patients must not have had any CLL-directed anticancer therapy within 5 half- lives of the therapy prior to Cycle 1 Day 1.
* Patients who have received a live vaccine within 30 days of planned start of study therapy. With regards to other type of vaccines, including SARS-Co2 vaccines, these are allowed.
* Patients requiring ongoing treatment with chronic high dose immunosuppressants (e.g., cyclosporine) or systemic steroids > 20 mg prednisone (or equivalent) QD. For example, patients with uncontrolled autoimmune haemolytic anaemia (AIHA) or idiopathic thrombocytopenia purpura (ITP), which requires > 20 mg once daily (QD) of prednisone (or equivalent) to maintain haemoglobin levels of >8.0 g/dL or platelets > 10,000 mL without transfusion support.
* History of transformation of CLL to aggressive non-Hodgkin lymphoma (Richter´s transformation or pro-lymphocytic leukaemia) which may otherwise interfere with the interpretation of the outcome of the study (including biomarker evaluation).
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia or fatigue. Any irAEs from prior immunotherapy must have complete resolution and must have resolved at least 2 weeks before Cycle1 Day1.
* Participants who are receiving any other investigational agents for this condition.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to roginolisib or venetoclax or their formulation components or prior anti- CD20 targeting agents more than 6 months before initiating study treatments.
* Patients with a history of systemic autoimmune disease.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A are ineligible. Moderate CYP3A inhibitors and P-gp inhibitors can be administered when venetoclax dose is reduced to 50%. Otherwise, venetoclax is contraindicated in patients requiring strong or moderate CYP3A inducers.

  * Because of ongoing research, regularly consulting medical reference databases is recommended. One such reference is the Website of the US-FDA: (Drug Interactions | Relevant Regulatory Guidance and Policy Documents | FDA)
  * As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Pregnant women are excluded from this study because venetoclax has the potential to cause embryo-fetal harm, and the potential for teratogenic or abortifacient effects with roginolisib is currently unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with roginolisib or venetoclax breastfeeding should be discontinued if the mother is treated with these agents.
* Patients with a history of other primary malignancy are excluded when they require therapy that will interfere with the investigational treatments. Exceptions are if the natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen. For example:

  * Malignancies surgically treated with curative intent and with no known active disease present for ≥2 years before the first dose of study treatment.
  * Adequately treated nonmelanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Surgically/adequately treated low-grade, early-stage, localized prostate cancer without evidence of disease or low risk localized prostate cancer on observation.
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
* History or presence of cardiovascular disease, which in the Investigator's opinion may impact the clinical trial participation. Patients with a QTcF > 470 msec at screening.
* History of tuberculosis treatment within the preceding two years.
* Ongoing systemic bacterial, fungal, or viral infections (including also hepatitis viral infection) at the time of initiation of study treatment (defined as requiring intravenous [IV] antimicrobial, antifungal or antiviral agents). Subjects on antimicrobial, antifungal or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met, there is no evidence of active infection at enrollment, and ongoing treatment does not have a significant risk of drug-drug interaction with venetoclax.
* Known Human immunodeficiency virus (HIV) infection which is treated with agents that can interfere with venetoclax due to potential drug-drug interactions or increased risk of myelotoxicity.
* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy.
* Known alcohol or substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Undetectable Minimal Residual Disease(uMRD) rate by ClonoSEQ assay | 1 year
  uMRD rate is defined as the proportion of participants with uMRD after treatment with either roginolisib plus venetoclax + rituximab, or venetoclax+ rituximab, as measured in bone marrow at a level of 10-4 by the clonoSEQ assay.

SECONDARY OUTCOMES:
Adverse Event of Interest Rate | 1 year
  Adverse event of interest rate is defined as the percentage of participants who experienced an adverse event including transaminitis, rash, diarrhea, colitis and pneumonitis as well as febrile neutropenia and infection. Assessment will be based on NCI CTCAE grading for non-hematologic toxicity, and iwCLL criteria for hematologic toxicity.
Undetectable Minimal Residual Disease(uMRD) rate by flow cytometry | 5 years
  uMRD as measured in blood at same timepoint as ClonoSeq.
Median Progression Free Survival(PFS) | 5 years
  PFS based on Kaplan Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation.
Median Overall Survival (OS) | 5 years
  Overall survival based on the Kaplan-Meier method is defined as the time from randomization to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Overall Response Rate (ORR) | 1 year
  ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) on treatment based on iwCLL criteria.
Duration of Response (DOR) | 5 years
  DOR is defined as the time from date of first documented confirmed objective response to date of first documented progressive disease (PD).
Complete Response Rate (CRR) | 1 year
  CRR was defined as the percentage of participants achieving complete response (CR) on treatment based on iwCLL criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu